CLINICAL TRIAL: NCT05545345
Title: Adjuvant Adenoidectomy Plus Tympanostomy Tube Placement for the Treatment of Chronic OME in Children
Brief Title: Adjuvant Adenoidectomy for the Treatment of Chronic OME in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-AdOME
Record Dates: First submitted 2022-08-04; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Otitis Media With Effusion in Children
Keywords: Otitis media with effusion; tympanostomy tube placement; adjuvant adenoidectomy; hearing outcome
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Adenoidectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TT (Active Comparator): Participants only receive tympanostomy tube placement.
  Interventions: Procedure: tympanostomy tube placement
- Ad+TT (Experimental): Participants will receive tympanostomy tube placement and concurrent adenoidectomy.
  Interventions: Procedure: tympanostomy tube placement; Procedure: adenoidectomy

INTERVENTIONS:
Procedure: tympanostomy tube placement — An incision will be made in the the tympanic membrane, through which a ventilation tube will be inserted.
Procedure: adenoidectomy — The adenoid is resected transorally under a 70° endoscope with microdebrider or coblator until torus tubarius and choanae are completely revealed.
  Arms: Ad+TT

SUMMARY:
This study aims to verify the efficacy of adjuvant adenoidectomy for children with chronic OME who become candidates for tympanostomy tube placement, and explore potential factors associated with the efficacy of adjuvant adenoidectomy.

DETAILED DESCRIPTION:
Otitis media with effusion is a common condition in children, and tympanostomy tube placement is the first-line treatment for those who requires surgical interventions. Adenoidectomy proves to be helpful to children over 4 years old, but the risks of adjuvant surgery is believed to somehow offset its benefits. This study is meant to verify if concurrent adenoidectomy provides extra benefits in resolving MEE, reducing AOM, and improving hearing and patients' quality of life to children who become candidates for TT.

ELIGIBILITY:
Inclusion Criteria:

* 1. Children 4-12 years of age.
* 2. Diagnosed with chronic OME. Diagnostic criteria: I. Middle ear effusion detected by otoscopy; II. Type B or C tympanograms; III. Symptoms/signs of OME persisted for >3 months;
* 3. Documented hearing loss ≥20dB (average threshold of 500Hz, 1000Hz and 2kHz in pure tone audiometry).
* 4. Adenoid hypertrophy (A/N ratio> 0.5 in lateral radiography of the nasopharynx).
* 5. Informed consent given by the patients and their guardians.

Exclusion Criteria:

1. Cleft palate or other systemic disorders.
2. Patients are diagnosed with other nose, sinuses or ear diseases that are eligible for surgical treatment.
3. Patients are diagnosed with OSAHS, tonsil hypertrophy ≥II° or scheduled for tonsillectomy.
4. History of tympanostomy tube placement.
5. Infection of the upper respiratory tract or acute rhinosinusitis over the past 7 days.
6. Sensorineural hearing loss.
7. Other situations that the investigators find unsuitable for the trial.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 380 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 1 year after tube removal
  Rate of OME recurrence
Rate of repeated tube placement | 1 year after tube removal
  proportion of patients who need repeated tube insertion

SECONDARY OUTCOMES:
AOM attacks | 1 year after tube removal
  The number of acute otitis media attacks
Otorrhea | 2 years after tube insertion
  Rate of Otorrhea
Pure tone audiometry | 2 years after tube insertion
  Change of pure tone audiometry thresholds compared with baseline
Otitis Media-6 and Pediatric Sleep Questionnaire | 2 years after tube insertion
  Change of questionnaire score. Otitis Media-6 score ranges from 6 to 42, and higher scores mean worse outcomes. Pediatric Sleep Questionnaire score ranges from 0 to 22, and higher scores mean worse outcomes.
Complications | 2 years after tube insertion
  Complications related to interventions of this study
Costs of OME-related visits and treatment | Through study completion, an average of 2 years
  Medical expenses associated with OME